CLINICAL TRIAL: NCT04366063
Title: Mesenchymal Stem Cell Therapy for Acute Respiratory Distress Syndrome in Coronavirus Infection: A Phase 2-3 Clinical Trial
Brief Title: Mesenchymal Stem Cell Therapy for SARS-CoV-2-related Acute Respiratory Distress Syndrome
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Royan Institute (Other Government)
Collaborators: Tehran University of Medical Sciences (Other); Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 991919; IRCT20200217046526N2 (Registry Identifier: Iranian Registry of Clinical Trials (IRCT))
Record Dates: First submitted 2020-04-20; First posted 2020-04-28 (Actual); Last update posted 2020-04-30 (Actual); Status verified 2020-04

CONDITIONS: Covid-19
Keywords: COVID-19; Acute Respiratory Distress Syndrome; 2019 Novel Coronavirus Pneumonia
MeSH Terms: conditions — COVID-19; Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Two MSC infusion (Experimental): Intervention Group1(n=20). Patients will receive two doses of MSCs 100×10e6 (±10%) intravenously plus Conventional treatment.
  Interventions: Biological: Cell therapy protocol 1
- Two MSC infusion Plus two EVs infusion (Experimental): Intervention Group 2 (n=20). Patients will receive two doses of MSCs 100×10e6 (±10%), intravenously plus two doses of EVs plus Conventional treatment
  Interventions: Biological: Cell therapy protocol 2
- Control (No Intervention): Control (n=20). Patients will conventional therapy for virus treatment and supportive care for ARDS will be used as control.

INTERVENTIONS:
Biological: Cell therapy protocol 1 — Cell therapy protocol 1(n=20). Patients will receive two doses of MSCs 100×10e6 (±10%) at Day 0 and Day 2 plus Conventional treatment.
  Arms: Two MSC infusion
Biological: Cell therapy protocol 2 — Patients will receive two doses of MSCs 100×10e6 (±10%)at Day 0 and Day 2, intravenously plus two doses of EVs at Day 4 and Day 6 plus conventional treatment.
  Arms: Two MSC infusion Plus two EVs infusion

SUMMARY:
Acute Respiratory Distress Syndrome (ARDS) is the major cause of death in the COVID-19 pandemic. In this trial, the safety and efficacy of Mesenchymal Stem Cells (MSC) for the treatment of ARDS in COVID-19 patients will be assessed.

DETAILED DESCRIPTION:
Acute respiratory distress syndrome (ARDS) is the major cause of death in the COVID 19 infection pandemic. It is a devastating clinical condition, caused by an acute and diffuse lung injury that requires management in the intensive care unit. It is caused by uncontrolled inflammation that leads to severe pulmonary alveolar damage and capillary membrane leakage, and progressive respiratory failure. There is no effective treatment for ARDS and the only supportive care strategies are the mainstay of therapy. Mesenchymal stem cells (MSCs) have high regenerative and immunomodulatory capacities. In preclinical research, ARDS, MSCs modulate the inflammatory response, augment tissue repair, enhance pathogen clearance, and reduce the severity of the injury, pulmonary dysfunction, and apoptosis. Moreover, many studies have shown that the anti-inflammatory effects of MSCs can significantly reduce virus (e.g., Influenza)-induced lung injury and mortality in animals. Since 2014 clinical trials are using MSC from variable sources [bone marrow (BM), fat, and umbilical cord (UC)] in the treatment of ARDS. Some of the clinical trials are ongoing and the final reports are not reported. In all final reports, the safety of the application of MSC has been documented and most of them implied improvement in mortality and decrease of morbidity. Moreover, experimental studies have demonstrated that MSCs or their extracellular vesicles (MSCs-EVs) significantly reduced lung inflammation and pathological impairment resulting from different types of lung injury. Also, macrophage phagocytosis, bacterial killing, and the outcome are improved. It is highly likely that MSCs-EVs have the same therapeutic effect on inoculation pneumonia as MSCs themselves.

Critically ill coronavirus documented cases suspicious to ARDS (mild or moderate) will be enrolled in the study. Our previous experiment (IRCT20200217046526N1) showed the safety of 3 injections of MSCs in patients with COVID-19. This multi-center trial will recruit 60 patients. All patients in all groups will receive conventional therapy for virus treatment and supportive care for ARDS.

The patients allocated randomly to three groups:

Control (n=20). Patients will conventional therapy for virus treatment and supportive care for ARDS will be used as control.

Intervention Group1 (n=20). Patients will receive two doses of MSCs 100×10e6 (±10%), at Day 0 and Day 2 intravenously.

Intervention Group 2 (n=20). Patients will receive two doses of MSCs 100×10e6 (±10%), at Day 0 and Day 2 plus two doses of extracellular vesicles (EVs) on Day 4 and Day 6 intravenously.

The clinical symptoms, pulmonary imaging, side effects, 28-days mortality inflammatory factors, etc. will be evaluated during the 28 days follow up.

ELIGIBILITY:
Inclusion Criteria:

* Confirmation of 2019-nCoV infection by RT-PCR
* Diagnosis of ARDS according to the Berlin definition of ARDS
* Requiring supplemental oxygen
* Pneumonia that is judged by chest radiograph or CT
* PaO2/oxygen absorption concentration (FiO2) ≤ 300MMHG
* Pulmonary imaging shows that the focused progress > 50% in 24-48 hours
* Mild to Moderate 2019-nCoV pneumonia/ stay in the ICU <48 hours
* SOFA score between 2-3 point

Exclusion Criteria:

* Severe allergies or allergies after 1st injection to stem cell preparations and their components
* Patients with a malignant tumor, other serious systemic diseases, and psychosis
* Co-Infection of HIV, tuberculosis, influenza virus, adenovirus, and other respiratory infection viruses
* Patients with a previous history of pulmonary embolism
* Be thought by researchers to be inappropriate to participate in this clinical study (Expected deaths within 48 hours, uncontrolled infections)
* Liver or kidney SOFA score of more than 3 points; combined with other organ failures (need organ support), Stage 4 severe chronic kidney disease or requiring dialysis (i.e. estimated glomerular filtration rate (eGFR) < 30)
* Pulmonary obstructive pneumonia, severe pulmonary interstitial fibrosis, alveolar proteinosis, allergic alveolitis, and other known viral pneumonia or bacterial pneumonia
* Continuous use of immunosuppressive agents or organ transplants in the past 6 months
* In vitro life support (ECMO, ECCO2R, RRT)
* Pregnant or lactating women
* Uncontrolled underlying disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-04-05 (Actual); Primary Completion 2020-06-06 (Estimated); Study Completion 2020-12-10 (Estimated)

PRIMARY OUTCOMES:
Adverse events assessment | From baseline to day 28
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0
Blood oxygen saturation | From baseline to day 14
  Evaluation of Pneumonia Improvement

SECONDARY OUTCOMES:
Intensive care unit-free days | Up to day 8
  Number of days
Clinical symptoms | From baseline to day 14
  Improvement of clinical symptoms including duration of fever, respiratory distress, pneumonia, cough, sneezing
Respiratory efficacy | From baseline to day 7
  increase in PaO2/FiO2 ratio from baseline to day 7
Biomarkers concentrations in plasma | At baseline, 7, 14, 28 days after the first intervention
  Biochemical examination

CONTACTS AND LOCATIONS:
Overall Officials: Abdol Hossein Shahverdi, Study Chair — Royan Institute; Hossein Baharvand, Professor, Principal Investigator — Department of Stem Cells Biology and Technology, Cell Science Research Center, Royan Institute for Stem Cells Biology & Technology, Iran
Locations (1):
- Royan Institute, Tehran, Iran

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR
Time Frame: 6 months after publication
Access Criteria: Researchers and clinicians